CLINICAL TRIAL: NCT05859256
Title: Efficacy of a Flossing Protocol and Manual Therapy in the Clinical and Functional Improvement of Young Subjects With Recurrent Ankle Sprains. A Randomized Clinical Study.
Brief Title: Flossing Protocol and Manual Therapy in Young Subjects With Recurrent Ankle Sprains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Flossing
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-05

CONDITIONS: Young People

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All evaluations will be carried out by one evaluator, blinded to the study conditions and the assignment of the players to the two study groups.
  In the subjects included in the control group, the same procedures will be carried out, but placing the flossing without tension and performing the Kaltenborn manual techniques without slipping and without joint mobilization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention consists of the application of a treatment protocol based on an initial active warm-up consisting of 3 active exercises, walking for 1 minute performing slow and controlled movement of the ankle, raising the heels, 15 repetitions, dorsiflexion of the ankle in the standing position. gentleman, 15 reps. Subsequently, the floss band will be placed, performing again the 3 active warm-up exercises with the band on. After this, the passive manual techniques will be carried out for the remaining time, removing the flossing at the end of the latter, and actively mobilizing again.
  Interventions: Other: Experimental
- Control group (Placebo Comparator): The subjects included in the control group will perform the same procedures, but placing the flossing without tension and performing the Kaltenborn manual techniques without sliding and without joint mobilization.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — The intervention consists of the application of a treatment protocol based on an initial active warm-up consisting of 3 active exercises, walking for 1 minute performing slow and controlled movement of the ankle, raising the heels, 15 repetitions, dorsiflexion of the ankle in the standing position. gentleman, 15 reps. Subsequently, the floss band will be placed, performing again the 3 active warm-up exercises with the band on. After this, the passive manual techniques will be carried out for the remaining time, removing the flossing at the end of the latter, and actively mobilizing again.
  Arms: Experimental group
Other: Control — The same procedures will be carried out, but placing the flossing without tension and performing the Kaltenborn manual techniques without sliding and without joint mobilization.
  Arms: Control group

SUMMARY:
The most frequent lateral ankle sprain mechanism consists of talocrural plantarflexion added to a subtalar inversion. The anterior talofibular ligament, in plantar flexion, suffers maximum stress, being very sensitive to injury mechanisms with inversion of the foot, being the cause of up to 70% of sprains. The risk of injury recurrence must be taken into account. In sports practice, this percentage of recurrence is especially relevant.

Randomized clinical study. Participants will be randomized to a control or experimental group. The dependent variable will be the range of motion in ankle dorsiflexion. Secondary variables will be pressure pain threshold, and stability of the foot and ankle. Three evaluations will be carried out: before the start of the study (T0), after the intervention (T1) and after a 4-week follow-up period (T2). All evaluations will be performed by one evaluator, blinded to player assignment The intervention consists of the application of a treatment protocol based on an initial active warm-up consisting of 3 active exercises, walking for 1 minute performing slow and controlled movement of the ankle, raising the heels, 15 repetitions, dorsiflexion of the ankle in the standing position. gentleman, 15 reps. Subsequently, the floss band will be placed, performing again the 3 active warm-up exercises with the band on. After this, the passive manual techniques will be carried out for the remaining time, removing the flossing at the end of the latter, and actively mobilizing again.

ELIGIBILITY:
Inclusion Criteria:

* Young people between 18 and 22 years old
* Who have suffered a previous sprain
* No chronic or degenerative musculoskeletal pathologies of the ankle or knee
* That they do physical activity regularly.

Exclusion Criteria:

* Have suffered a sprain in the last 6 months
* Being receiving another physiotherapy treatment at the time of the study
* Not signing the informed consent document.

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-05-06 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline ankle range of motion after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  Using an analog goniometer, range of motion was measured. This instrument has shown excellent reliability. The joint range in plantar and dorsiflexion was measured. The unit of measurement is degrees (the higher the degree, the greater the mobility).

SECONDARY OUTCOMES:
Change from baseline pressure pain threshold treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  Pressure pain threshold will be measured with a pressure algometer (Wagner FDIX model, Wagner Instruments, CT, USA). Pressure will be progressively applied until the sensation begins to be painful. Pressure pain threshold will be measured bilaterally in the region ventral to the lateral malleolus.
Change from baseline foot and ankle stability after treatment and at 4 weeks | Screening visit, within the first seven days after treatment and after four weeks follow-up
  The biomechanical analysis of gait and balance will be evaluated using an Rs Scan® pressure platform and a FootScan® pressure measurement system. This scientific version biomechanical examination device measures plantar pressure using an X-Y array of resistive pressure sensitive sensors that are sequentially scanned. The system records pressure data when the subject is standing or walking on the platform. The measurements will be made with the basic platform of 0.5m with 4096 sensors with resistive technology and 300Hz data acquisition frequency. The biomechanics of gait will be analyzed with the analysis of the probes and the static balance in a time of 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Study Director — Universidad de Oviedo
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided